CLINICAL TRIAL: NCT06531915
Title: Comparison of Efficacy and Safety Between Ciprofol and Remimazolam During Fiberoptic Bronchoscopy: a Study Protocol for a Single-center, Double-blind, Randomized Controlled Trial
Brief Title: Comparison of Efficacy and Safety Between Ciprofol and Remimazolam During Fiberoptic Bronchoscopy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Fiberoptic bronchoscopy
Record Dates: First submitted 2024-05-21; First posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-05

CONDITIONS: Fiberoptic Bronchoscopy
MeSH Terms: interventions — (2-(1R)-1-cyclopropyl)ethyl-6-isopropyl-phenol; remimazolam

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ciprofol group (Experimental)
  Interventions: Drug: Ciprofol
- Remimazolam group (Active Comparator)
  Interventions: Drug: Remimazolam

INTERVENTIONS:
Drug: Ciprofol — Participants in the ciprofol group will be intravenously injected with 0.4 mg/kg of ciprofol (batch number H20200013, Haisike Pharmaceutical Co., Ltd., Liaoning, China) and sufentanil (0.2 μg/kg).
  Arms: Ciprofol group
Drug: Remimazolam — Participants in the remimazolam group will be intravenously injected with 0.1 mg/kg of remimazolam besylate (batch number HR7056, Hengrui Pharmaceutical Co., Ltd., Jiangsu, China) and sufentanil (0.2 μg/kg).
  Arms: Remimazolam group

SUMMARY:
Both ciprofol and remimazolam have been found to be potential alternatives to propofol (a commonly used anesthesia) during fiberoptic bronchoscopy, while the efficacy and safety between ciprofol and remimazolam have not been reported. This study aims to compare the efficacy and safety between ciprofol and remimazolam in patients undergoing fiberoptic bronchoscopy.

ELIGIBILITY:
Inclusion Criteria:

1. male or female patients with age ≥ 18 years old;
2. scheduled to undergo bronchoscopy under laryngeal mask airway;
3. with American Society of Anesthesiologists (ASA) physical status classes II to Ⅲ; and
4. volunteering to participate in this study and signing an informed consent form.

Exclusion Criteria:

1. with contraindications to deep sedation/general anesthesia or with a history of sedation/anesthesia accidents;
2. allergic to eggs, bean products, or experimental drugs (ciprofol, sufentanil, or remimazolam);
3. difficult airway;
4. with bradycardia or other serious cardiovascular diseases;
5. with severe damages or diseases in important organs such as the lungs, brain, liver, or kidneys;
6. using sedatives or antidepressants for a long time;
7. pregnant or lactating women; and (8) unable to communicate or cooperate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
The success rate of fiberoptic bronchoscopy | 24 hours after fiberoptic bronchoscopy

SECONDARY OUTCOMES:
Induction time | 24 hours after fiberoptic bronchoscopy
Procedure time | 24 hours after fiberoptic bronchoscopy
Awake time | 24 hours after fiberoptic bronchoscopy
Recovery time | 24 hours after fiberoptic bronchoscopy
Stay time in PACU | 24 hours after fiberoptic bronchoscopy
Supplemental times of experimental drugs (ciprofol or remimazolam) | 24 hours after fiberoptic bronchoscopy
Doses of experimental drugs (ciprofol or remimazolam) | 24 hours after fiberoptic bronchoscopy
Times of using rescue sedative drug | 24 hours after fiberoptic bronchoscopy
Doses of using rescue sedative drug | 24 hours after fiberoptic bronchoscopy
Incidence of adverse events | 24 hours after fiberoptic bronchoscopy
Patients' satisfaction | 24 hours after fiberoptic bronchoscopy
  Patients' satisfaction is assessed using the Satisfaction Scale reported by Luo et al. The Satisfaction Scale ranges from 0 to 10 points and contains five items. The higher score indicates better satisfaction.
Heart rate | 6 minutes after fiberoptic bronchoscopy
SBP | 6 minutes after fiberoptic bronchoscopy
Diastolic blood pressure | 6 minutes after fiberoptic bronchoscopy
SpO2 | 6 minutes after fiberoptic bronchoscopy

IPD SHARING:
Plan to Share IPD: No